CLINICAL TRIAL: NCT06796673
Title: Retina BioBank: Retina Biomarkers for a Deeper Understanding of Vitreoretinal and Systemic Diseases
Acronym: RBBK
Status: Enrolling by invitation | Type: Observational
Sponsor: Greater Houston Retina Research (Other)
Responsible Party: Sponsor
Other Study IDs: RBBK
Record Dates: First submitted 2023-02-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Other Retinal Disorders; Retinal Disease; Retinal Vascular Disorder
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Aqueous humor, vitreous humor, intraoperative tissue, and/or saliva will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RBBK study is a non-interventional, prospective study that will characterize disease state biomarker levels from aqueous humor, vitreous humor, intraoperative tissue and saliva of subjects with various retinal and systemic pathologies.

DETAILED DESCRIPTION:
The RBBK study is a non-interventional, prospective study that will characterize disease state biomarker levels from aqueous humor, vitreous humor, intraoperative tissue and saliva of subjects with various retinal and systemic pathologies.

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Men or women > 18 years of age
2. Subjects with vitreoretinal disease in at least one eye receiving a retinal treatment intervention
3. Able and willing to provide signed informed consent

The study will consist of a single visit and a retrospective chart review. The study visit will consist of:

1. Screening for eligibility;
2. Aqueous humor collection (if applicable);
3. Vitreous humor collection (if applicable);
4. Intraoperative tissue (if applicable); and
5. Saliva collection

If applicable, approximately 50 microliters (or more, up to 1000 microliters) of aqueous fluid will be collected by anterior chamber paracentesis according to standard clinical procedures. If applicable, up to 2 milliliters of vitreous fluid will be collected according to standard clinical procedures. Specific tissue, such as scar tissue, are routinely removed from the eye during vitreoretinal procedures. When being removed during a standard of care surgical procedure, these tissues may be collected. Saliva will also be collected according to instructions found in the Saliva Oragene Dx Collection Kit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with vitreoretinal disease in at least one eye receiving a retinal treatment intervention

Exclusion Criteria:

1. Prior intraocular or subtenon steroid injection in the study eye within the prior 1 month of signing informed consent
2. Intraocular or refractive surgery in the study eye within 30 days of signing informed consent
3. Systemic anti-VEGF treatment within 90 days of signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retina Consultants of Texas patient population.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
To quantify levels of disease state biomarkers implicated in the pathogenesis of various retinal and systemic pathologies | Baseline
  An analysis of the ocular fluids and tissues of patients with various vitreoretinal diseases would allow for the development of a deeper understanding of the processes that contribute to their onset and may ultimately provide insight in methods to refine treatment and management options.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C. Wykoff, MD, PhD, Principal Investigator — Greater Houston Retina Research
Locations (3):
- United States (3):
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Mesquida M, Drawnel F, Fauser S. The role of inflammation in diabetic eye disease. Semin Immunopathol. 2019 Jul;41(4):427-445. doi: 10.1007/s00281-019-00750-7. Epub 2019 Jun 7. PMID 31175392
- [Background] Mesquita J, Castro-de-Sousa JP, Vaz-Pereira S, Neves A, Passarinha LA, Tomaz CT. Evaluation of the growth factors VEGF-a and VEGF-B in the vitreous and serum of patients with macular and retinal vascular diseases. Growth Factors. 2018 Apr;36(1-2):48-57. doi: 10.1080/08977194.2018.1477140. Epub 2018 Jul 3. PMID 29969324
- [Background] Amadio M, Govoni S, Pascale A. Targeting VEGF in eye neovascularization: What's new?: A comprehensive review on current therapies and oligonucleotide-based interventions under development. Pharmacol Res. 2016 Jan;103:253-69. doi: 10.1016/j.phrs.2015.11.027. Epub 2015 Dec 8. PMID 26678602
- [Background] Witmer AN, Vrensen GF, Van Noorden CJ, Schlingemann RO. Vascular endothelial growth factors and angiogenesis in eye disease. Prog Retin Eye Res. 2003 Jan;22(1):1-29. doi: 10.1016/s1350-9462(02)00043-5. PMID 12597922
- [Background] Zhang X, Bao S, Lai D, Rapkins RW, Gillies MC. Intravitreal triamcinolone acetonide inhibits breakdown of the blood-retinal barrier through differential regulation of VEGF-A and its receptors in early diabetic rat retinas. Diabetes. 2008 Apr;57(4):1026-33. doi: 10.2337/db07-0982. Epub 2008 Jan 3. PMID 18174522
- [Background] Hofman P, Blaauwgeers HG, Tolentino MJ, Adamis AP, Nunes Cardozo BJ, Vrensen GF, Schlingemann RO. VEGF-A induced hyperpermeability of blood-retinal barrier endothelium in vivo is predominantly associated with pinocytotic vesicular transport and not with formation of fenestrations. Vascular endothelial growth factor-A. Curr Eye Res. 2000 Aug;21(2):637-45. PMID 11148600
- [Background] Wu H, Hwang DK, Song X, Tao Y. Association between Aqueous Cytokines and Diabetic Retinopathy Stage. J Ophthalmol. 2017;2017:9402198. doi: 10.1155/2017/9402198. Epub 2017 Jun 7. PMID 28680705
- [Background] Dong N, Xu B, Wang B, Chu L. Study of 27 aqueous humor cytokines in patients with type 2 diabetes with or without retinopathy. Mol Vis. 2013 Aug 4;19:1734-46. Print 2013. PMID 23922491
- [Background] Kersten E, Paun CC, Schellevis RL, Hoyng CB, Delcourt C, Lengyel I, Peto T, Ueffing M, Klaver CCW, Dammeier S, den Hollander AI, de Jong EK. Systemic and ocular fluid compounds as potential biomarkers in age-related macular degeneration. Surv Ophthalmol. 2018 Jan-Feb;63(1):9-39. doi: 10.1016/j.survophthal.2017.05.003. Epub 2017 May 15. PMID 28522341
- [Background] Knickelbein JE, Chan CC, Sen HN, Ferris FL, Nussenblatt RB. Inflammatory Mechanisms of Age-related Macular Degeneration. Int Ophthalmol Clin. 2015 Summer;55(3):63-78. doi: 10.1097/IIO.0000000000000073. No abstract available. PMID 26035762
- [Background] Jonas JB, Tao Y, Neumaier M, Findeisen P. Cytokine concentration in aqueous humour of eyes with exudative age-related macular degeneration. Acta Ophthalmol. 2012 Aug;90(5):e381-8. doi: 10.1111/j.1755-3768.2012.02414.x. Epub 2012 Apr 10. PMID 22490043
- [Background] Park KS, Kim JW, An JH, Woo JM. Elevated plasma pentraxin 3 and its association with retinal vein occlusion. Korean J Ophthalmol. 2014 Dec;28(6):460-5. doi: 10.3341/kjo.2014.28.6.460. Epub 2014 Nov 19. PMID 25435748
- [Background] Noma H, Funatsu H, Yamasaki M, Tsukamoto H, Mimura T, Sone T, Hirayama T, Tamura H, Yamashita H, Minamoto A, Mishima HK. Aqueous humour levels of cytokines are correlated to vitreous levels and severity of macular oedema in branch retinal vein occlusion. Eye (Lond). 2008 Jan;22(1):42-8. doi: 10.1038/sj.eye.6702498. Epub 2006 Jul 7. PMID 16826241
- [Background] Lopez-Contreras AK, Martinez-Ruiz MG, Olvera-Montano C, Robles-Rivera RR, Arevalo-Simental DE, Castellanos-Gonzalez JA, Hernandez-Chavez A, Huerta-Olvera SG, Cardona-Munoz EG, Rodriguez-Carrizalez AD. Importance of the Use of Oxidative Stress Biomarkers and Inflammatory Profile in Aqueous and Vitreous Humor in Diabetic Retinopathy. Antioxidants (Basel). 2020 Sep 20;9(9):891. doi: 10.3390/antiox9090891. PMID 32962301